CLINICAL TRIAL: NCT07387757
Title: Effectiveness of a Physical Therapy Intervention Using Exergames in Mental Health
Brief Title: Exergames in Mental Health
Acronym: PHYSIOGAME
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Inés Llamas-Ramos, Principal Investigator, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: MENTALHEALTH2026
Record Dates: First submitted 2026-01-17; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Mental Disorders
Keywords: Exergames; Physiotherapy; Exercise
MeSH Terms: conditions — Mental Disorders; Motor Activity | interventions — Exercise; Dosage Forms; Exergaming; Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exergames (Experimental): Participants will undergo physical therapy based on active video games using the Nintendo Switch, with games selected for their ability to promote physical activity:
  * Ring Fit Adventure (guided training, integrated breathing).
  * Nintendo Switch Sports (overall movement, coordination).
  * Just Dance (motivational cardiovascular activation).
  Interventions: Other: Control
- Conventional (Active Comparator): This group will continue to carry out the usual intervention
  Interventions: Procedure: EXERCISE TRAINING WITH OR WITHOUT MEDICATION

INTERVENTIONS:
Procedure: EXERCISE TRAINING WITH OR WITHOUT MEDICATION — Participants will undergo physical therapy based on active video games using the Nintendo Switch, with games selected for their ability to promote physical activity, for 2 sessions/week, 40 minutes, for 4 weeks:
  * Ring Fit Adventure (guided training, integrated breathing).
  * Nintendo Switch Sports (overall movement, coordination).
  * Just Dance (motivational cardiovascular activation).
  Other Names: Exergames with Nintendo Switch
  Arms: Conventional
Other: Control — This group will continue to perform the usual intervention that has scheduled.
  Other Names: Control group
  Arms: Exergames

SUMMARY:
Mental health and stress-related disorders have a growing impact on physical functioning, motivation, and participation in daily activities. Several studies indicate that integrating physical therapy into mental health programs improves functional status, reduces associated physical symptoms (fatigue, muscle tension, somatization), and promotes emotional regulation through movement. However, its implementation in clinical services remains limited. This project proposes to evaluate the effectiveness of an innovative mental health-oriented physical therapy program using active video games (exergames) on the Nintendo Switch platform, an accessible, motivating tool that can be adapted to each patient's functional level.

Objective: To determine whether a structured physiotherapy program based on exergames promotes physical exercise, improves quality of life, and increases therapeutic adherence in patients with mental illness.

Methods: An experimental pilot study will be conducted, implementing an intervention over 4 weeks, with 2 sessions per week lasting 40 minutes. Participants (n=12) will be assigned to an intervention group (exergames with Nintendo Switch) or a control group (usual routine). Quality of life, motivation, and therapeutic adherence will be assessed using the World Health Organization Quality of Life - BREF (WHOQOL-BREF) questionnaire, the Intrinsic Motivation Inventory, and a satisfaction questionnaire.

Expected results: The intervention group is expected to show better quality of life, greater motivation to exercise, and greater adherence to treatment. It is also expected to demonstrate that exergames are a viable tool, accepted by patients and incorporable into mental health physical therapy programs.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 65 years of age.
* Clinical diagnosis of mental illness.
* Psychopharmacological stability for at least 4 weeks prior to enrollment.
* Ability to perform light-moderate physical exercise.
* Written informed consent.

Exclusion Criteria:

* Severe psychiatric diagnoses with psychotic involvement or high suicide risk.
* Neurological or musculoskeletal conditions that limit the safe practice of exercise.
* Active substance use that interferes with the intervention.
* Moderate-severe cognitive impairment.
* Recent participation (<3 months) in other intervention studies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life: World Health Organization Quality of Life - BREF (WHOQOL-BREF) | Day 1, day 15 and day 29
  The WHOQOL-BREF is a questionnaire developed by the World Health Organization to assess perceived quality of life. It is an abbreviated version of the WHOQOL-100 and contains 26 items that explore four main dimensions: physical health, psychological health, social relationships, and environment. It also includes two general questions on the overall perception of quality of life and satisfaction with health. It is a widely used, valid, and reliable instrument in different populations, providing a comprehensive and comparative view of people's well-being in their life context. It has been used in psychiatric populations and in studies with people with various mental disorders, and there is scientific evidence of its use and psychometric properties in this context.

SECONDARY OUTCOMES:
Motivation: Intrinsic Motivation Inventory (IMI) | Day 1, day 15 and day 29
  The Intrinsic Motivation Inventory (IMI) is a questionnaire designed to assess the degree of intrinsic motivation a person experiences when performing a specific activity. It measures key psychological factors related to motivation, such as interest/enjoyment, perceived competence, effort, perceived value or usefulness of the task, pressure/stress, and experience of choice or autonomy. It is a widely used tool in studies of motivation, learning, and adherence to intervention programs, as it provides insight into which aspects of an activity promote participant engagement and persistence. The IMI has also been used in psychiatric populations and in studies related to mental health.
Adverse effects | Day 1, day 15 and day 29
  Self-diary

CONTACTS AND LOCATIONS:
Locations (1):
- University of Salamanca, Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No